CLINICAL TRIAL: NCT04189562
Title: A Text Messaging (SMS) Intervention to Improve Adherence to Stimulant Medications in Children With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief of the Clinical and Research Programs in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-P-002715
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Attention Deficit/Hyperactivity Disorder; ADHD; SMS Intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMS Intervention (Experimental): All parents of participants will receive customized text messages once a day, Sunday through Friday, for a duration of 9 months that will include reminders to adhere to the individualized medication regimen, reminders to call their clinician for a prescription refill followed by reminders to pick up medication from the pharmacy, and educational reminders about ADHD and its treatment.
  Interventions: Other: SMS Intervention

INTERVENTIONS:
Other: SMS Intervention — Delivery of text messages will use the text messaging program Simple Online Family Intervention for ADHD (SOFIA).

SUMMARY:
This study will assess the efficacy of the text messaging (SMS-based) disease management intervention for children with Attention Deficit/Hyperactivity Disorder (ADHD) using the timeliness of stimulant prescription renewals over a 9-month period.

Parents of participants in the study will receive customized text messages once a day, Sunday through Friday, for a duration of 9 months. The text messages will include reminders to adhere to the individualized medication regimen, reminders to call their child's clinician for a prescription refill followed by reminders to pick up medication from the pharmacy, and educational reminders about ADHD and its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-12 years of age of both sexes and their parent
* A diagnosis of ICD-10 or DSM 5 diagnosis of Attention Deficit/Hyperactivity Disorder including the following ICD codes (F90 Attention-deficit hyperactivity disorders; F90.0 Attention-deficit hyperactivity disorder, predominantly inattentive type; F90.1 Attention- deficit hyperactivity disorder, predominantly hyperactive type; F90.2 Attention-deficit hyperactivity disorder, combined type;F90.8 Attention-deficit hyperactivity disorder, other type; F90.9 Attention-deficit hyperactivity disorder, unspecified type) and/or the following DSM 5 diagnoses (314.01, F90.2 Attention-deficit/hyperactivity disorder, combined presentation; 314.01, F90.1 Attention-deficit/hyperactivity disorder, predominantly hyperactive/impulsive presentation;314.00, F90.0 Attention- deficit/hyperactivity disorder, predominantly inattentive presentation)
* Starting or currently on stimulant medication including (Amphetamine/Dextroamphetamine (Adderall);Dextroamphetamine (Dexedrine, ProCentra, Zenzedi, Adderall XR); Dexmethylphenidate (Focalin, Focalin XR); Methylphenidate (Ritalin, Ritalin SR, Metadate ER, Methylin ER, Concerta, Daytrana, Metadate CD, Quillivant XR, Ritalin LA); Amphetamine sulfate (Evekeo); Lisdexamfetamine (Vyvanse))
* Proficient in English
* Has a cellular phone with text messaging capabilities and is interested in and willing to receive free of charge text messages

Exclusion Criteria:

* Investigator and his/her immediate family
* Unwilling/unable to comply with study procedures

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Adherence to Stimulants | 9 months
  Adherence will be analyzed using the timeliness of stimulant medication prescription renewals over the 9 month period as documented in the participants medical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No